CLINICAL TRIAL: NCT07192926
Title: The Impact of Sarcopenia and CRP-TyG Index (CTI) on Immunotherapy Response in Patients With Metastatic Non-Small Cell Lung Cancer: A Single-Center Retrospective Analysis
Brief Title: Sarcopenia and CRP-TyG Index (CTI) as Predictors of Immunotherapy Response in Metastatic Non-Small Cell Lung Cancer
Acronym: SARCO-CTI
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncologist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK2-2025-452; AEŞH-BADEK2-2025-452 (Other: Ankara Etlik City Hospital Scientific Research Ethics Committee)
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Non-small Cell Lung Cancer; Neoplasm
Keywords: sarcopenia; CTI Score; Immunotherapy; Immune Checkpoint Inhibitors; PD-1 / PD-L1 Inhibitors; Prognostic Biomarker; Survival Outcomes; Skeletal Muscle Index (SMI); CRP-TyG Index (CTI)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Sarcopenia; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Immune Checkpoint Inhibitors; Nivolumab; pembrolizumab; atezolizumab; durvalumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic NSCLC Patients Treated With Immunotherapy: This cohort includes 115 adult patients with histologically confirmed metastatic non-small cell lung cancer (mNSCLC) who received immune checkpoint inhibitors at Ankara Etlik City Hospital between November 2022 and December 2024. Patients had available baseline and 3-month CT imaging for sarcopenia assessment and laboratory data for CRP, triglycerides, and fasting glucose to calculate the CRP-TyG Index (CTI).
  Interventions: Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Drug: Immune Checkpoint Inhibitors — Retrospective analysis of patients with metastatic non-small cell lung cancer (mNSCLC) who received standard-of-care immune checkpoint inhibitors, including PD-1 and PD-L1 inhibitors (e.g., nivolumab, pembrolizumab, atezolizumab, durvalumab). Patients received these agents as part of routine clinical practice; no experimental intervention was administered in this study.
  Other Names: Nivolumab; Pembrolizumab; Atezolizumab; Durvalumab

SUMMARY:
This study investigates the impact of sarcopenia and the CRP-TyG Index (CTI) on immunotherapy outcomes in patients with metastatic non-small cell lung cancer (NSCLC). Medical records of 115 adult patients treated with immune checkpoint inhibitors at Ankara Etlik City Hospital between November 2022 and December 2024 will be retrospectively analyzed.

Sarcopenia will be determined from CT-based skeletal muscle index (SMI) measurements at the L3 vertebral level. SMI will be calculated as skeletal muscle area (cm²) divided by height squared (m²), with sex-specific cut-offs (≤52.4 cm²/m² for men, ≤38.5 cm²/m² for women). CTI will be calculated from CRP, triglycerides, and fasting glucose values.

Primary outcome is objective response rate (ORR, RECIST 1.1). Secondary outcomes include 1-year progression-free survival (PFS), 1-year overall survival (OS), treatment duration, and adverse events (CTCAE v5.0).

DETAILED DESCRIPTION:
Metastatic non-small cell lung cancer (mNSCLC) is among the leading causes of cancer-related mortality worldwide. Immune checkpoint inhibitors (ICIs) targeting PD-1/PD-L1 have improved survival outcomes, yet responses remain heterogeneous. Prognostic biomarkers such as sarcopenia and systemic inflammation-metabolism indices may help optimize patient selection.

This retrospective, single-center cohort study will analyze 115 adult patients with mNSCLC treated with ICIs at Ankara Etlik City Hospital between November 2022 and December 2024. Sarcopenia will be assessed from computed tomography (CT) imaging at the L3 vertebral level by calculating skeletal muscle index (SMI = skeletal muscle area [cm²] / height² [m²]). Patients will be classified as sarcopenic if SMI ≤52.4 cm²/m² for men or ≤38.5 cm²/m² for women. Both baseline and 3-month CT scans will be analyzed to assess dynamic changes (ΔSMI).

The CRP-TyG Index (CTI) will be calculated as:

TyG = ln [triglycerides (mg/dL) × fasting glucose (mg/dL) / 2] CTI = 0.412 × ln [CRP (mg/L)] + TyG Patients will be categorized into low- and high-risk groups using the published cut-off of 4.78.

The primary endpoint is objective response rate (ORR, RECIST v1.1). Secondary endpoints include 12-month progression-free survival (PFS), overall survival (OS), treatment duration, adverse events (graded by CTCAE v5.0), and sarcopenia dynamics. Associations between CTI and sarcopenia will also be explored. Statistical analyses include multivariable logistic regression for ORR and Cox proportional hazards models for PFS/OS, adjusting for age, sex, and ECOG status.

This study aims to integrate radiological (sarcopenia), biochemical (CRP, triglycerides, glucose), and clinical outcomes to determine whether sarcopenia and CTI can serve as practical prognostic markers for immunotherapy in real-world mNSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histologically confirmed diagnosis of metastatic non-small cell lung cancer (mNSCLC).
* Received at least one cycle of immune checkpoint inhibitor (PD-1 or PD-L1 inhibitor) as part of routine clinical care.
* Availability of baseline CT imaging (within 4 weeks before treatment initiation) and follow-up CT imaging at approximately 3 months.
* Availability of baseline laboratory data including C-reactive protein (CRP), triglycerides, and fasting glucose.
* Adequate clinical records for evaluation of treatment response and survival outcomes.

Exclusion Criteria:

* Age <18 years.
* Patients without immunotherapy treatment.
* Incomplete or missing CT imaging or laboratory data required for sarcopenia or CTI assessment.
* Patients lost to follow-up before first radiological evaluation.
* Prior malignancy within 5 years (except adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population consists of 115 adult patients with histologically confirmed metastatic non-small cell lung cancer (mNSCLC) who received immune checkpoint inhibitors at Ankara Etlik City Hospital between November 2022 and December 2024. All included patients had available baseline and 3-month CT scans for sarcopenia assessment and laboratory data for calculation of the CRP-TyG Index (CTI).
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to 12 months after initiation of immunotherapy
  Proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST 1.1 criteria, based on radiological evaluation.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Baseline to 12 months
  Time from initiation of immunotherapy to disease progression or death from any cause, whichever occurs first.
Overall Survival (OS) | Baseline to 12 months
  Time from initiation of immunotherapy to death from any cause.
Treatment Duration | Baseline to end of treatment (up to 12 months)
  Duration of immunotherapy treatment, measured from initiation to discontinuation for any reason.
Adverse Events (Toxicity Profile) | Baseline to 12 months
  Incidence and severity of treatment-related adverse events, graded according to CTCAE version 5.0.
Sarcopenia Status at Baseline | At baseline (0 months)
  Skeletal Muscle Index (SMI = skeletal muscle area [cm²] / height² [m²]) measured at L3 level.
  Minimum value: near 0 (exceptionally low muscle mass) No theoretical maximum, but typical range: ~20-80 cm²/m² Lower values indicate worse muscle status. Cut-offs: ≤52.4 cm²/m² (men), ≤38.5 cm²/m² (women) define sarcopenia.
Sarcopenia Status at 3 Months | 3 months after initiation of immunotherapy
  Skeletal Muscle Index (SMI) at 3-month CT scan. SMI reassessed at ~3 months. Same cut-offs as above. Same cut-offs as baseline (≤52.4 cm²/m² for men, ≤38.5 cm²/m² for women).

OTHER OUTCOMES:
Change in Sarcopenia (ΔSMI) | Baseline to 3 months
  Difference in SMI between baseline and 3 months. Patients classified as stable/improved vs worsened.
CRP-TyG Index (CTI) Prognostic Value | At baseline (0 months)
  CTI calculated as: CTI = 0.412 × ln [CRP (mg/L)] + ln [Triglycerides (mg/dL) × Fasting Glucose (mg/dL) / 2].
  CTI is a continuous score with no absolute minimum/maximum; typically ranges 2-7.
  Higher CTI values indicate higher systemic inflammation-metabolic risk. Patients will be stratified at 4.78 (low risk vs. high risk).
Correlation Between Sarcopenia and CTI | Baseline to 12 months
  Relationship between baseline sarcopenia (SMI cut-offs) and baseline CTI (cut-off 4.78), and their combined effect on immunotherapy outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Galip Can Uyar, MD, Principal Investigator — Etlik City Hospital Medical Oncology Department
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik City Hospital Medical Oncology Department, Ankara, Yenimahalle
  - Etlik City Hospital Radiology Department, Ankara, Yenimahalle

IPD SHARING:
Plan to Share IPD: No